CLINICAL TRIAL: NCT06036563
Title: A Multicenter Prospective Diagnostic Test: Screening and Differentiating Common Cancers (Cancers of Lung, Stomach, Colorectum, Esophagus, Liver, Breast and Pancreas) Based on Peripheral Blood Cell-Free DNA Sequencing
Brief Title: Prospective Screening and Differentiating Common Cancers Using Peripheral Blood Cell-Free DNA Sequencing
Status: Recruiting | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Tang-Du Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); First Hospital of China Medical University (Other); People's Hospital of Ningxia Hui Autonomous Region (Other); Xinjiang Medical University (Other); Guanxian People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Other Study IDs: KY20232260-F-1
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cancer Diagnosis; LungCancer; Gastric Cancer; Liver Cancer; Colorectal Cancer; Esophagus Cancer; Breast Cancer; Pancreas Cancer
Keywords: multicancer screening; liquid biopsy; cell-free DNA; methylation; machine learning
MeSH Terms: conditions — Stomach Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Breast Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — 15~20ml peripheral venous blood sample from each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multicenter prospective cancer-screening cohort: The cohort, including cancer patients and non-cancer patients, will be prospectively enrolled in from different departments and centers. The focused cancers include lung cancer, gastric cancer, colorectal cancer, liver cancer, esophagus cancer, breast cancer and pancreas cancer.

SUMMARY:
The goal of this observational study is to screen and differentiate common cancers in participants with or without suspicious lesions. The main question the investigators aim to answer is: Can the developed model, using peripheral blood cell-free DNA sequencing, work well in screening and classifying common cancers especially in the early stages? Participants will undergo the collection of 15~20ml of blood and 1~2 telephone follow-up calls.

ELIGIBILITY:
Inclusion Criteria:

1. >20 and < 80 years old.
2. Cancer group: Newly diagnosed cancer patients with a confirmed pathological diagnosis within 90 days before blood collection or within 30 days after blood collection, including lung cancer, esophageal cancer, breast cancer, stomach cancer, colorectal cancer, liver cancer, and pancreatic cancer.

Non-cancer group: Individuals who have not been diagnosed with cancer during routine physical examinations and one-year follow-up.

Exclusion Criteria:

1. Uncontrolled or active systemic diseases, such as autoimmune diseases, tuberculosis, AIDS, etc.
2. New onset, recurrence, or exacerbation of various inflammations within 2 weeks before blood collection, or the presence of fever, use of corticosteroids.
3. New onset or exacerbation of thromboembolic diseases, hemorrhagic diseases, or those who have received allogeneic blood transfusion within 1 month before blood collection.
4. Any cancer treatment performed within the past 3 years.
5. Individuals who have undergone organ or bone marrow transplantation.
6. Participants during pregnancy or lactation.
7. Individuals with malnutrition, severe mental illness, or genetic diseases.
8. Other diseases or conditions deemed by the physician as unsuitable for participation in this study.
9. Individuals who are unable to sign an informed consent form.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PASS 21.0 is used to calculate the sample size for diagnostic tests. Based on the specificity and sensitivity of different cancer diagnoses in current and reported studies, the specificity is preset at 98%, and the sensitivity is preset at 75%. A two-sided test is chosen, with a confidence level of 1-α=0.9, and a confidence interval width of 10%. The minimum sample size for the diagnostic test is calculated as follows: each type of cancer should have no less than 202 cases in the diagnostic test, and the total number of cancer subjects should not be less than 1414. The ratio of cancer subjects to non-cancer subjects is set at 1:1. Considering the possibility of loss to follow-up, unqualified sample quality, and dropout during the study, the sample size for this study is preset at 3200.
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | Immediately after test completion
  This refers to the ability of the test (peripheral blood cell-free DNA sequencing) to correctly classify individuals into the categories of having or not having the disease. It is a measure of the test's overall effectiveness. The reference test is histological test for cancers or one-year follow-up for non-cancers.
sensitivity | Immediately after test completion
  This is the ability of the test (peripheral blood cell-free DNA sequencing) to correctly identify those with the disease. It is the proportion of true positive results (those with the disease who test positive) to the total number of individuals who actually have the disease. The reference test is histological test for cancers or one-year follow-up for non-cancers.
specificity | Immediately after test completion
  This is the ability of the test (peripheral blood cell-free DNA sequencing) to correctly identify those without disease. It is the proportion of true negative results (those without the disease who test negative) to the total number of individuals who actually do not have the disease. The reference test is histological test for cancers or one-year follow-up for non-cancers.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - First Affiliated Hospital of Air Force Military Medical University, Xi'an, Shaanxi
  - Tang-du Hospital, Xi'an, Shaanxi
  - Guanxian People's Hospital, Liaocheng, Shandong
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nikanjam M, Kato S, Kurzrock R. Liquid biopsy: current technology and clinical applications. J Hematol Oncol. 2022 Sep 12;15(1):131. doi: 10.1186/s13045-022-01351-y. PMID 36096847
- [Background] Gao Q, Lin YP, Li BS, Wang GQ, Dong LQ, Shen BY, Lou WH, Wu WC, Ge D, Zhu QL, Xu Y, Xu JM, Chang WJ, Lan P, Zhou PH, He MJ, Qiao GB, Chuai SK, Zang RY, Shi TY, Tan LJ, Yin J, Zeng Q, Su XF, Wang ZD, Zhao XQ, Nian WQ, Zhang S, Zhou J, Cai SL, Zhang ZH, Fan J. Unintrusive multi-cancer detection by circulating cell-free DNA methylation sequencing (THUNDER): development and independent validation studies. Ann Oncol. 2023 May;34(5):486-495. doi: 10.1016/j.annonc.2023.02.010. Epub 2023 Feb 26. PMID 36849097
- [Background] Jamshidi A, Liu MC, Klein EA, Venn O, Hubbell E, Beausang JF, Gross S, Melton C, Fields AP, Liu Q, Zhang N, Fung ET, Kurtzman KN, Amini H, Betts C, Civello D, Freese P, Calef R, Davydov K, Fayzullina S, Hou C, Jiang R, Jung B, Tang S, Demas V, Newman J, Sakarya O, Scott E, Shenoy A, Shojaee S, Steffen KK, Nicula V, Chien TC, Bagaria S, Hunkapiller N, Desai M, Dong Z, Richards DA, Yeatman TJ, Cohn AL, Thiel DD, Berry DA, Tummala MK, McIntyre K, Sekeres MA, Bryce A, Aravanis AM, Seiden MV, Swanton C. Evaluation of cell-free DNA approaches for multi-cancer early detection. Cancer Cell. 2022 Dec 12;40(12):1537-1549.e12. doi: 10.1016/j.ccell.2022.10.022. Epub 2022 Nov 17. PMID 36400018
- [Background] Helzer KT, Sharifi MN, Sperger JM, Shi Y, Annala M, Bootsma ML, Reese SR, Taylor A, Kaufmann KR, Krause HK, Schehr JL, Sethakorn N, Kosoff D, Kyriakopoulos C, Burkard ME, Rydzewski NR, Yu M, Harari PM, Bassetti M, Blitzer G, Floberg J, Sjostrom M, Quigley DA, Dehm SM, Armstrong AJ, Beltran H, McKay RR, Feng FY, O'Regan R, Wisinski KB, Emamekhoo H, Wyatt AW, Lang JM, Zhao SG. Fragmentomic analysis of circulating tumor DNA-targeted cancer panels. Ann Oncol. 2023 Sep;34(9):813-825. doi: 10.1016/j.annonc.2023.06.001. Epub 2023 Jun 16. PMID 37330052
- [Background] Fan R, Chen L, Zhao S, Yang H, Li Z, Qian Y, Ma H, Liu X, Wang C, Liang X, Bai J, Xie J, Fan X, Xie Q, Hao X, Wang C, Yang S, Gao Y, Bai H, Dou X, Liu J, Wu L, Jiang G, Xia Q, Zheng D, Rao H, Xia J, Shang J, Gao P, Xie D, Yu Y, Yang Y, Gao H, Liu Y, Sun A, Jiang Y, Yu Y, Niu J, Sun J, Wang H, Hou J. Novel, high accuracy models for hepatocellular carcinoma prediction based on longitudinal data and cell-free DNA signatures. J Hepatol. 2023 Oct;79(4):933-944. doi: 10.1016/j.jhep.2023.05.039. Epub 2023 Jun 10. PMID 37302583